CLINICAL TRIAL: NCT03333980
Title: A Non-interventional Observational Clinical Study to Document the Clinical Course of Patients 12 Months or More Following an Ischaemic Stroke
Brief Title: An Ischaemic Stroke Observational Study
Status: Completed | Type: Observational
Sponsor: ReNeuron Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: RN-CS-0002
Record Dates: First submitted 2017-09-26; First posted 2017-11-07 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A non-interventional observational clinical study to document the clinical course of patients at 12 months or more following an ischaemic stroke

DETAILED DESCRIPTION:
Primary objective:

To document and better define the prognostic characteristics of residual disability 12 months or more following an ischaemic stroke in patients that originally participated in the preceding clinical study RN-CS-0001.

Other objective:

To inform the design of efficient Phase 2/3 studies when screening potentially efficacious interventions for signals of activity which merit further development.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to give informed consent or witnessed informed consent in the event that the patient is unable to sign informed consent due to physical impairments.
* Participation in the preceding study RN-CS-0001
* Completion of at least one of the 4 functional assessment tests (ARAT, BI, NIHSS, mRS) at any time point on the previous study RN-CS-0001
* Ability to participate in all assessments and attend all visits

Exclusion Criteria:

* Any additional incidence of stroke (Ischaemic or Haemorrhagic) since participation in the previous study RN-CS-0001 (since the last CS-0001 assessment visit date).
* Incidence of significant other disease that judged by the investigator would confound completion of all functional assessments (not excluding patients that can complete at least one functional assessment with no confounding factor from significant other disease).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients assessed as part of the preceding study RN-CS-0001 which forms the list of potential patients for this study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Compare functional assessment scores collected in this study with the preceding RN-CS-0001 study | 12-months
  Compare functional assessment scores collected in RN-CS-0002 with the preceding RN-CS-0001 study to better understand stroke symptom recovery and progress

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - New Queen Elizabeth Hospital, Birmingham
  - Ninewells Hospital & Medical School, Dundee
  - Queen Elizabeth University Hospital., Glasgow
  - University College London Hospital Stroke Research Centre, London
  - The University of Manchester Institute of Cardiovascular Research, Manchester
  - Nottingham City Hospital, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton